CLINICAL TRIAL: NCT04119778
Title: Improving Sleep in Lung Cancer Patients: A Randomized Controlled Trial of Aerobic Exercise and Tai-chi Interventions
Brief Title: Improving Sleep in Lung Cancer Patients: A Trial of Aerobic Exercise and Tai-chi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Chia-Chin Lin, Professor and Head, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW18154，; HKECCREC-2019-014 (Registry Identifier: Hong Kong East Cluster Research Ethics Committee); KC/KE-19-0039/ER-3 (Registry Identifier: Research Ethics Committee (Kowloon Central/Kowloon East))
Record Dates: First submitted 2019-09-06; First posted 2019-10-08 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Sleep
MeSH Terms: interventions — Exercise; Tai Ji

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise (Experimental): The exercise intervention will last 16 weeks, comprised of home-based exercise with weekly telephone counselling to encourage participants to continue to exercise, supplemented with 8 supervised exercise sessions (2 sessions per month). Each session will last for an hour. The supervised exercise sessions will be provided by professional exercise specialists twice in the first week in each month throughout the intervention period, an hour each time. Exercise trainers will lead the classes. Each class will include both aerobic exercise and resistance exercise. They are encouraged to do aerobic exercise for at least 150 min weekly at a moderate intensity level, as well as perform resistance exercises alternate day. Participants are also provided an exercise diary, containing details of their weekly prescribed exercises and the scales they have to refer to.
  Interventions: Behavioral: Aerobic Exercise, Tai chi
- Tai chi (Experimental): Our tai-chi classes will be based on a 16-form tai-chi exercise set. The classes will run twice a week for 16 weeks with each session lasting approximately 60 minutes. Classes will be taught by an experienced tai-chi master, who will explain the theory behind tai-chi and the principles of the techniques. The supervised session includes a warm up, self-massage and a guided run through of the movements, breathing techniques, and relaxation in tai-chi. The tai-chi master will guide participants to practice the tai-chi they learn in the classes at home each day. Upon completion of the 16 weeks course, participants will be encouraged to continue their tai-chi practice, given guidance on local services and programmes they may join if they wish to.
  Interventions: Behavioral: Aerobic Exercise, Tai chi
- Self Management Group (No Intervention): Participants randomised to the control group shall receive written information on health levels of physical activity, which they can participate in at home (self-management) and continue to receive their usual care, participants will be followed up with an assessment at 16 weeks and one year. At the end of the evaluation stage of the study, survivors in the control group will be invited to take part in an intervention of their choice.

INTERVENTIONS:
Behavioral: Aerobic Exercise, Tai chi — They are aerobic and mind-body exercise respectively.
  Arms: Aerobic Exercise; Tai chi

SUMMARY:
Lung cancer is one of the commonest cancers around the world. Sleep disturbances are commonly reported by lung cancer patients. Meanwhile, disturbed sleep is associated with several health problems, including shortened survival period. Thus, lung cancer imposes a substantial health burden on patients and society both locally and world widely. On top of the classical clinical therapies, additional approaches that could result in improved sleep are needed.

Previous studies, including our own, have shown that physical exercise, such as aerobic walking, improves lung cancer patient's physical fitness particularly cardiovascular fitness, circadian rhythm and immune function. Another popular mode of exercise in Chinese population is tai-chi. With emphasis on breathing and concentration, tai-chi exhibits extra benefits for stress-relieving and psychological well-being. Those benefits of exercise have long been implicated for better sleep of cancer patients. The promising benefits of aerobic exercise or tai-chi, as non-pharmacological interventions, urge for need of rigorous evidence on the effectiveness of these interventions in improving sleep outcomes. However, to date, there has been no report from a randomized controlled trial (RCT) to study the effect of aerobic exercise or tai-chi on sleep of lung cancer patients.

This proposed research is designed to conduct a three-arm RCT comparing aerobic exercise, tai-chi to usual care in non-small cell lung cancer patients. Recruited participants will be randomised into three groups: 1) a 16-week aerobic exercise group, 2) a 16-week tai-chi program group, and 3) a self-management control group. Aerobic exercise and tai-chi program will be conducted by certificated coaches. Life-long adherence to the practice in intervention groups is encouraged.

Through this project, the investigators aim to evaluate if 1) aerobic exercise or 2) tai-chi intervention promote subjective sleep quality in lung cancer patients compared to control, as the primary outcome of this study. The investigators shall also examine if tai-chi practice can provide similar improvement in sleep quality compared with ordinary exercise. Using biomarkers including circadian rhythm, cardio-respiratory fitness, further provides objective measures for bio-physiological effectiveness of the interventions. The associations of those biological measures and psycho-social status with sleep outcomes will be further explored.

Findings of this study will provide crucial information on the evidence-based practice by physical exercise or tai-chi to improve sleep of lung cancer patients. This study will also have far-reaching significance in providing important scientific evidence to policymakers to integrate physical activity into routine clinical management as an add-on treatment for lung cancer patients in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed of stage IIIB, or IV non-small-cell lung cancer confirmed by pathology
2. Patients are not currently engaged in other research or participant in any other exercise or mind-body classes
3. Patients aged 18 years old, or above
4. Patients who can communicate in Cantonese, Mandarin
5. Patients with no other cancer diagnosis within the previous 1 year
6. Patients report not doing regular exercises (defined <150 min of moderate-intensity exercise weekly) in daily living, but are able to attend either exercise or tai-chi classes at scheduled times
7. Patients with ECOG 0-1
8. Patients being conscious and alert.
9. Patients who can read and write in Chinese

Exclusion Criteria:

* Patients suffering from a diagnosed active neurological, substance abuse and /or psychiatric disorders (i.e. depression, chronic insomnia)。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Quality of Sleep (Subjective)- Pittsburgh Sleep Quality Index | 1 year
  To assess the change of quality of sleep, the Chinese version of the Pittsburgh Sleep Quality Index, from baseline at 16-week and 1 year

SECONDARY OUTCOMES:
Levels of physical activity | Baseline, 16-week, 1 year
  To measure compliance to exercise all participants will be measured for their level of physical activity in daily living. Physical activity will be quantified with a non-invasive small-size wrist-worn piezoelectric accelerometer (Actigraph; Ambulatory Monitoring Inc., New York). Actigraphy has been shown to provide valid assessments of physical activity. The user-defined time interval for the count of wrist accelerations is 1 min. Patients will be asked to wear the actigraph for at least 3 consecutive 24-hour spans. Each patient will keep a diary for times of rising and retiring.
Circadian rhythms- cortisol rhythms | Baseline, and 1 year
  We will measure circadian rhythms using biomarkers that have been linked to survival of cancer patients, cortisol rhythms will be measured using saliva samples collected before and after intervention. The cortisol levels will be measured using enzyme-linked immunosorbent assay (ELISA) kits. The saliva will be collected using Salivettes at following time points: 0.5 hour, 4 hour, 8 hour and 12 hour after habitual wake time (referred as circadian time).
Circadian rhythms- melatonin rhythms | Baseline, and 1 year
  We will measure circadian rhythms using biomarkers that have been linked to survival of cancer patients, melatonin rhythms will be measured using saliva samples collected before and after intervention. The melatonin levels will be measured using enzyme-linked immunosorbent assay (ELISA) kits. The saliva will be collected using Salivettes at following time points: 0.5 hour, 4 hour, 8 hour and 12 hour after habitual wake time (referred as circadian time).
Cardio-respiratory fitness- 6-minute walking test | Baseline, 16-week, 1 year
  Cardio-respiratory fitness shall be evaluated using the 6-minute walking test (6MWT). The 6MWT has been widely used to assess cardio-respiratory fitness in lung cancer patients [28-30]. The 6MWT requires participants to walk on an even and flat surface between two cones set 30m apart, with the object being the participant walking as far as possible within the 6 minutes period (if participant cannot continue for the 6 minutes, the test will end). The walking test is measured in units of meters walked at the end of the 6 minutes.
Physical functioning- Get Active Questionnaire | Baseline, 16-week, 1 year
  Physical fitness will a be assessed using the Get Active Questionnaire (GAQ). The GAQ assesses if participants are safe to participate in the interventions and ensures if participants can perform the exercises within the intervention.
Physical functioning- timed up and go test | Baseline, 16-week, 1 year
  This test evaluates participants' agility.
Physical functioning-sit to stand test | Baseline, 16-week, 1 year
  This test evaluates participants' muscle strength.
Physical functioning- single leg standing test | Baseline, 16-week, 1 year
  This test evaluates participants' balance.
Immune functions- cytotoxic activity of natural killer (NK) cells, and spontaneous or phytohemagglutinin (PHA)-stimulated T-lymphocyte proliferation | Baseline, 1 year
  For each participant, 10 ml of peripheral blood will be collected before and after intervention in intervention groups, as well as in control group at the same time points, for some immune functional studies. The peripheral blood mononuclear cells are isolated for measurements of immune functions. Immune functions will be analyzed by cytotoxic activity of natural killer (NK) cells, and spontaneous or phytohemagglutinin (PHA)-stimulated T-lymphocyte proliferation.
Health-related quality of Life- European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire | Baseline, 16-week, 1 year
  Health related QoL is an important outcome for lung cancer patients and plays an important impact on prognosis. The Chinese version of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30). It will be evaluated by three parts, global score, symptom score and functional score with the range of 0-100. Higher score in global and functional aspects denote better quality of life while lower score in symptom aspects denotes better quality of life.
Health-related quality of Life- European Organization for Research and Treatment of Cancer Quality of Life Core corresponding lung cancer-specific module | Baseline, 16-week, 1 year
  Health related QoL is an important outcome for lung cancer patients and plays an important impact on prognosis. The Chinese version of the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire corresponding lung cancer-specific module (QLQ-LC13) shall be used as measurements of QoL. Lower score denotes better quality of life. The range of score is 0-100.
Psychological Distress- Hospital Anxiety and Depression Score | Baseline, 16-week, 1 year
  To evaluate psychological distress the Hospital Anxiety and Depression Score (HADS) will be used. The HADS comprises seven items each for anxiety and depression. Each item of the anxiety subscale and the depression subscale was scored on a 4-point scale. This scale is a reliable tool, and is widely used to assess patients with cancer.
Fatigue- Brief Fatigue Inventory | Baseline, 16-week, 1 year
  Fatigue will be measured by the Chinese version of the Brief Fatigue Inventory (BFI). The BFI was developed to measure fatigue in cancer patients. It consists of 9 items with each item scored on a 0-10 scale. The BFI measures patients' fatigue when symptoms are at their worst, least, usual and currently during the normal waking hours, with 0 indicating no fatigue, and 10 being fatigue as bad as one can imagine. Other items include fatigues interaction with patients' general activity, mood, waking ability, normal work (includes both work outside the home and housework), relations with other people, ability to think clearly, and enjoyment of life. The interference is measured with 0 being does not interfere, and 10 being completely interferes.
Quality of Sleep (Objective)- Actigraph | Baseline, 16-week, 1 year
  Actigraph will serve as an objective measure for assessing sleep parameters, such as sleep efficiency, total sleep time.
Fried frailty Criteria | Baseline, 16-week, 1 year
  Frailty will be measured by weight loss, exhaustion, low physical activity, slowness and weakness.
One-year survival rate | 1 year
  One-year relative survival rate will be retrieved from patients' medical record.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Takemura N, Cheung DST, Fong DYT, Lee AWM, Lam TC, Ho JC, Kam TY, Chik JYK, Lin CC. Comparative effect of Tai Chi and aerobic exercise on cognitive function in advanced lung cancer survivors with perceived cognitive impairment: a three-arm randomized controlled trial with mediation analysis. J Cancer Surviv. 2025 Dec;19(6):1938-1947. doi: 10.1007/s11764-024-01607-1. Epub 2024 May 1. PMID 38691272
- [Derived] Takemura N, Cheung DST, Fong DYT, Lee AWM, Lam TC, Ho JC, Kam TY, Chik JYK, Lin CC. Effectiveness of Aerobic Exercise and Tai Chi Interventions on Sleep Quality in Patients With Advanced Lung Cancer: A Randomized Clinical Trial. JAMA Oncol. 2024 Feb 1;10(2):176-184. doi: 10.1001/jamaoncol.2023.5248. PMID 38060250
- [Derived] Takemura N, Cheung DST, Fong DYT, Lee AWM, Lam TC, Ho JC, Kam TY, Chik JYK, Lin CC. Relationship of subjective and objective sleep measures with physical performance in advanced-stage lung cancer patients. Sci Rep. 2021 Aug 26;11(1):17208. doi: 10.1038/s41598-021-96481-7. PMID 34446756